CLINICAL TRIAL: NCT01975441
Title: Evaluate Triple-Drug Therapy With Diethylcarbamize (DEC), Albendazole (ALB) and Ivermectin (IVM) That Could Accelerate LF Elimination Outside of Africa
Brief Title: Eval 3-Drug Therapy Diethylcarbamize, Albendazole and Ivermectin That Could Accelerate LF Elimination Outside of Africa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Christopher L. King, MD, PhD, Professor/PI, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CWRU 3 vs 2 LF ELIM PNG
Record Dates: First submitted 2013-10-28; First posted 2013-11-04 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Lymphatic Filariasis
Keywords: Diethycarbamazine; Albendazole; Ivermectin; Lymphatic filariasis
MeSH Terms: conditions — Elephantiasis, Filarial | interventions — Diethylcarbamazine; Albendazole; Albumins; Ivermectin; Intravital Microscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- standard treatment (Active Comparator): Diethylcarbamazine 6 mg/kg + Albendazole 400 mg administered annually (at 0, 12, and 24 months).
  Interventions: Drug: Diethylcarbamazine; Drug: Albendazole
- DEC 6 mg/kg + Alb 400 mg x 1 (Experimental): Diethylcarbamazine 6 mg/kg + Albendazole 400 mg given once
  Interventions: Drug: Diethylcarbamazine; Drug: Albendazole
- DEC + ALB + IVM (Experimental): Diethylcarbamazine 6 mg/kg + Albendazole 400 mg + Ivermectin 200 µg/kg administered once only at the beginning of the RCT (0 month)
  Interventions: Drug: Diethylcarbamazine; Drug: Albendazole; Drug: Ivermectin

INTERVENTIONS:
Drug: Diethylcarbamazine — Diethylcarbamazine 6mg/kg
  Other Names: DEC
Drug: Albendazole — Albendazole 400mg
  Other Names: ALB, Albenda
Drug: Ivermectin — Ivermectin 200 mcg/kg
  Other Names: IVM, Stromectol
  Arms: DEC + ALB + IVM

SUMMARY:
This study will determine if a combination of 3 drugs used to treat the infection that cause lymphatic filariasis (LF) due to Wuchereria bancrofti infection are more effective in killing or sterilizing the adult worms compared to just 2 of the 3 drugs that usually given to treat this infection. The three drugs used together are called albendazole (ALB), ivermectin (IVM) and diethylcarbamazine (DEC). The usual treatment in Papua New Guinea (PNG) for lymphatic filariasis are DEC and ALB. A combination of these 3 drugs has not been previously used to treat LF.

DETAILED DESCRIPTION:
This study will determine whether a single dose of the triple drug regimen of DEC/Iver/Alb is non-inferior to annual treatments with DEC/Alb in inducing sustained clearance of Mf in LF infected subjects (>50 Mf/ml) at 36 months post-treatment. This study also tests the hypothesis that single dose of triple drug is super in sustained clearance of microfilariae compared to single dose of DEC/ALB.

There will be 3 treatment arms as follows:

1. The comparator (standard treatment) DEC 6 mg/kg + Alb 400 mg administered annually (at 0, 12, and 24 months).
2. DEC 6 mg/kg + Alb 400 mg given once
3. DEC 6 mg/kg + Alb 400 mg + Iver 200 µg/kg administered once only at the beginning of the RCT (0 month).

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18-65 years
* >50 mf/ml in finger stick blood samples
* Willing to give informed consent

Exclusion Criteria:

* Prior treatment for LF within last 5 years
* Pregnant (do pregnancy test)
* Hemoglobin < 7 g/dl
* permanent disability, serious medical illness that prevents or impedes study participation and/or comprehension
* AST/ALT and creatinine > 1.5 upper limit of normal.
* Urine dipstick with glucose ≥ 2+ and/or protein ≥ 2+

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with total clearance of in Wuchereria bancrofti (Wb) microfilaria (mf) | at 36 months

SECONDARY OUTCOMES:
Percentage of subjects with total clearance of Mf at 24 months. | 24 months
Percent reduction in W. bancrofti antigen levels compared to baseline measured at 24 and 36 months | 24 months and 36 months
Percent of subjects who become circulating antigen negative at 24 months and 36 months after the beginning of the study | 24 months and 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter Siba, PhD, Principal Investigator — Papua New Guinea Institution for Medical Research
Locations (1):
- Papua New Guinean Institute for Medical Research, Maprik, East Sepik Province, Papua New Guinea

REFERENCES:
- [Derived] King CL, Suamani J, Sanuku N, Cheng YC, Satofan S, Mancuso B, Goss CW, Robinson LJ, Siba PM, Weil GJ, Kazura JW. A Trial of a Triple-Drug Treatment for Lymphatic Filariasis. N Engl J Med. 2018 Nov 8;379(19):1801-1810. doi: 10.1056/NEJMoa1706854. PMID 30403937
- [Derived] Thomsen EK, Sanuku N, Baea M, Satofan S, Maki E, Lombore B, Schmidt MS, Siba PM, Weil GJ, Kazura JW, Fleckenstein LL, King CL. Efficacy, Safety, and Pharmacokinetics of Coadministered Diethylcarbamazine, Albendazole, and Ivermectin for Treatment of Bancroftian Filariasis. Clin Infect Dis. 2016 Feb 1;62(3):334-341. doi: 10.1093/cid/civ882. Epub 2015 Oct 20. PMID 26486704